CLINICAL TRIAL: NCT05408663
Title: EXT608 in Human Healthy Adults; A First-in-Human, Randomized, Double-Blind, Placebo-controlled, Single Dose Escalation Study
Brief Title: A Phase 1 Study of EXT608 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Extend Biosciences Inc. (Industry)
Collaborators: Integrated Medical Development (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EXT608-101; R44DK107231 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Safety Issues
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Single ascending dose with up to 6 sequential dose escalation cohorts. Participants will be randomized to either study intervention (EXT608) or placebo
Who Masked: Participant, Investigator
Masking Description: Double (Participant, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental- EXT608 (Experimental): Up to 6 sequential dose escalation cohorts will receive a single dose of EXT608 administered as a subcutaneous injection
  Interventions: Drug: EXT608
- Placebo comparator (Placebo Comparator): Up to 6 participants will receive matching placebo administered as a subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EXT608 — EXT608 is an investigational drug administered via subcutaneous injection
  Other Names: test drug
  Arms: Experimental- EXT608
Other: Placebo — matching placebo administered via subcutaneous injection
  Arms: Placebo comparator

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose safety and tolerability study of EXT608 in healthy subjects. There will be up to 6 sequential dose escalation cohorts of 4 participants. In each cohort 3 participants will receive EXT608 and 1 participant will receive placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, first-in-human, placebo-controlled single ascending dose study to study the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of EXT608 in healthy adult participants.

Participants will be enrolled into 1 of up to 6 planned single dose cohorts in ascending fashion.

Each cohort will consist of 4 participants randomized to receive either EXT608 or placebo, whereby 3 will receive a single injection of EXT608 and 1 will receive matching placebo.

Up to 6 dosing cohorts are planned with no single dose escalation to exceed a 3-fold dose increment. A Data Monitoring Board will review the seven-day safety data in each cohort before authorizing the initiation of the next cohort.

A screening visit will take place within 28 days of dosing. Eligible participants for each cohort will be admitted to the Clinical Research Unit (CRU) 1 day prior to dosing and remain in the CRU through at least 72 hours after dosing for safety and PK assessments before discharge. The total confinement period will be 4 nights, unless extended for management of Adverse Events (AEs) at the discretion of the Investigator

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 55 years of age.
2. Body mass index between 18.5 and 32 kilogram per square meter (kg/m2), inclusive, with a body weight greater than or equal to (>=) 45 kg.
3. In general good medical health with no clinically significant or relevant abnormalities,
4. A clinical safety laboratory parameter of hemoglobin greater than (>) 11.7 gram per deciliter (g/dl) (females) or 13.1 g/dl (males) and less than (<) 16 g/dl (females) or 17.4 g/dl (males) or, if out of this range, deemed not clinically significant by the Investigator.
5. Total serum calcium (Se-Ca) within laboratory normal limits.
6. Serum parathyroid hormone (PTH) concentration within normal laboratory limits.

Exclusion Criteria:

1. Evidence of clinically significant (CS) neurologic, cardiovascular, pulmonary, hepatic, hematopoietic disease, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, serious allergy, allergic skin rash, or psychiatric disorder
2. History of drug abuse
3. Currently using any medication including over-the-counter (OTC), herbal or homeopathic preparations
4. Pregnant, nursing, or planning a pregnancy during the course of or within 3 months of completing this study
5. History of cancer or other malignancy, with the exception of basal cell carcinoma that has been in remission for at least 5 years
6. Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or a human immunodeficiency virus (HIV)
7. Alanine transaminase (ALT) and/or aspartate transaminase (AST) >1.5 the upper limit of normal (ULN)
8. Increased baseline risk for osteosarcoma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hales, PhD, Study Director — Extend Biosciences
Locations (1):
- PRA, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Comparator: Six participants (one per cohort) received matching placebo administered as a subcutaneous injection
- Experimental- EXT608 4ug: Cohort 1: 4 ug Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 12 ug: Cohort 2: 12 ug Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 36 ug: Cohort 3: 36 ug Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 108 ug: Cohort 4: 108 ug Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 324 ug: Cohort 5: 324 ug Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 216 ug: Cohort 6: 216 ug Three participants received a single dose of EXT608 administered as a subcutaneous injection
Period: Overall Study
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12 ug | Experimental- EXT608 36 ug | Experimental- EXT608 108 ug | Experimental- EXT608 324 ug | Experimental- EXT608 216 ug
Started | 6 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 6 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental- EXT608 4ug; Experimental- EXT608 12 ug; Experimental- EXT608 36ug; Experimental- EXT608 108ug; Experimental- EXT608 324ug; Experimental- EXT608 216ug: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12 ug | Experimental- EXT608 36ug | Experimental- EXT608 108ug | Experimental- EXT608 324ug | Experimental- EXT608 216ug | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 3 | 2 | 2 | 13
  Male | 5 | 1 | 1 | 2 | 0 | 1 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 6 | 3 | 2 | 3 | 2 | 2 | 3 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 6
  White | 4 | 1 | 1 | 0 | 3 | 3 | 2 | 14
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Characterize the Safety and Tolerability of EXT608
Description: Incidence, nature and severity of adverse events (AEs) and withdrawals due to Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Day 0 to Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Comparator: Six participants (1 in each of 6 sequential dose escalation cohorts) received matching placebo administered as a subcutaneous injection
- Experimental - EXT608 4 ug: Cohort 1: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental - EXT608 12 ug: Cohort 2: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental - EXT608 36 ug: Cohort 3: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental - EXT608 108 ug: Cohort 4: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental - EXT608 324 ug: Cohort 5: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental - EXT608 216 ug: Cohort 6: Three participants received a single dose of EXT608 administered as a subcutaneous injection
Arm/Group | Placebo - Comparator | Experimental - EXT608 4 ug | Experimental - EXT608 12 ug | Experimental - EXT608 36 ug | Experimental - EXT608 108 ug | Experimental - EXT608 324 ug | Experimental - EXT608 216 ug
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  Adverse Event | 2 | 2 | 0 | 0 | 0 | 0 | 0
  Any AE That Might Be Related to Study Drug | 0 | 0 | 1 | 0 | 1 | 2 | 0
  Serious Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No Adverse Event | 4 | 1 | 2 | 3 | 2 | 1 | 3
  Withdrawal from Study | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Characterize the Safety and Tolerability of EXT608
Description: Frequency and severity of post-dose change from baseline of hematology, serum chemistry, urinalysis, electrocardiogram (ECG), vital signs and physical examination findings
Time Frame: Day 0 - Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Comparator: Six participants (1 participant in each of 6 sequential dose escalation cohorts) received matching placebo administered as a subcutaneous injection
- Experimental- EXT608 4ug: Cohort 1: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 12ug: Cohort 2: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 36ug: Cohort 3: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 108ug: Cohort 4: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 324ug: Cohort 5: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 216ug: Cohort 6: Three participants received a single dose of EXT608 administered as a subcutaneous injection
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12ug | Experimental- EXT608 36ug | Experimental- EXT608 108ug | Experimental- EXT608 324ug | Experimental- EXT608 216ug
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Characterize the Safety and Tolerability of EXT608
Description: Percentage of participants with injection or infusion site reactions - edema
Time Frame: Day 0 - Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Comparator: Six participants (1 in each of 6 sequential dose escalation cohorts) received matching placebo administered as a subcutaneous injection
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12ug | Experimental- EXT608 36ug | Experimental- EXT608 108ug | Experimental- EXT608 324ug | Experimental- EXT608 216ug
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Single Dose Pharmacokinetics (PK) - Area Under the Curve (AUC)
Description: Area under the curve
Time Frame: Day 0 to Day 7
Measure: Mean (Standard Deviation); unit: pg*Day/mL
Groups:
- Placebo Comparator: Six participants (one in each of 6 sequential dose escalation cohorts) received matching placebo administered as a subcutaneous injection
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12ug | Experimental- EXT608 36ug | Experimental- EXT608 108ug | Experimental- EXT608 324ug | Experimental- EXT608 216ug
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3
pg*Day/mL | NA (NA) — below the level of detection | NA (NA) — below the level of detection | NA (NA) — below the level of detection | 358.3 (119.2) | 1613 (379.3) | 4903 (475.7) | 2091 (794.3)

5. Secondary Outcome: Single Dose PK - Cmax
Description: Maximum observed concentration
Time Frame: 0-24 hr
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Experimental- EXT608 4ug: Cohort 1: Up to 3 participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 12ug: Cohort 2: Up to 3 participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 36ug: Cohort 3: Up to 3 participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 108ug: Cohort 4: Up to 3 participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 324ug: Cohort 5: Up to 3 participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 216ug: Cohort 6: Up to 3 participants received a single dose of EXT608 administered as a subcutaneous injection
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12ug | Experimental- EXT608 36ug | Experimental- EXT608 108ug | Experimental- EXT608 324ug | Experimental- EXT608 216ug
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3
pg/mL | NA (NA) — below the level of detection | NA (NA) — below the level of detection | NA (NA) — below the level of detection | 489.3 (271.1) | 1156 (339) | 4967 (1950) | 1266 (489.4)

6. Secondary Outcome: Single Dose PK - Tmax
Description: Time to reach maximum observed plasma concentration
Time Frame: Day 0 to Day 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Placebo Comparator | Experimental- EXT608 4ug | Experimental- EXT608 12ug | Experimental- EXT608 36ug | Experimental- EXT608 108ug | Experimental- EXT608 324ug | Experimental- EXT608 216ug
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 3
hr | NA (NA) — below the level of detection | NA (NA) — below the level of detection | NA (NA) — below the level of detection | 3.3 (1.15) | 5.3 (2.30) | 2.7 (1.16) | 4.0 (0.03)

ADVERSE EVENTS:
Time Frame: 28 days
Description: Adverse events were graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Groups:
- Experimental- EXT608 4 ug: Cohort 1: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 12 ug: Cohort 2: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 36 ug: Cohort 3: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 108 ug: Cohort 4: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 324 ug: Cohort 5: Three participants received a single dose of EXT608 administered as a subcutaneous injection
- Experimental- EXT608 216 ug: Cohort 7: Three participants received a single dose of EXT608 administered as a subcutaneous injection
Arm/Group | Placebo Comparator | Experimental- EXT608 4 ug | Experimental- EXT608 12 ug | Experimental- EXT608 36 ug | Experimental- EXT608 108 ug | Experimental- EXT608 324 ug | Experimental- EXT608 216 ug
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/6 | 2/3 | 1/3 | 0/3 | 2/3 | 2/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator (N=6) | Experimental- EXT608 4 ug (N=3) | Experimental- EXT608 12 ug (N=3) | Experimental- EXT608 36 ug (N=3) | Experimental- EXT608 108 ug (N=3) | Experimental- EXT608 324 ug (N=3) | Experimental- EXT608 216 ug (N=3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality Disclosure Agreement

DOCUMENTS (3):
  • Study Protocol (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT05408663/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05408663/SAP_001.pdf
  • Informed Consent Form (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT05408663/ICF_002.pdf